CLINICAL TRIAL: NCT02096913
Title: The Rho-Inhibitor Ibuprofen for the Treatment of Acute Spinal Cord Injury: Investigation of Safety, Feasibility and Pharmacokinetics
Brief Title: Safety Study of Ibuprofen to Treat Acute Traumatic Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jan M. Schwab, MD, PhD (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Sponsor-Investigator, Jan M. Schwab, MD, PhD, Prof. Dr. Dr., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ibuprofen-SCI-Safety; 2011-000584-28 (EudraCT Number)
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Injury
Keywords: Rho-Inhibition; Plasticity; Neurological Function; RhoA; Ibuprofen; NSAIDs
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dolormin® extra (Ibuprofen) 4 weeks (Active Comparator)
  Interventions: Drug: Dolormin® extra (Ibuprofen)
- Dolormin® extra (Ibuprofen) 12 weeks (Active Comparator)
  Interventions: Drug: Dolormin® extra (Ibuprofen)

INTERVENTIONS:
Drug: Dolormin® extra (Ibuprofen) — Ibuprofen Tablets (as lysine-salt) 2400mg/d (400mg 2-2-2) applied orally for 4 weeks (Arm I; n=6).
  In order to reduce the risk of damage to the gastrointestinal mucosa Pantoprazole is applied as concomitant medication in a dosage 40mg/d during the treatment period.
  Other Names: Ibuprofen-DL-Lysinsalz
  Arms: Dolormin® extra (Ibuprofen) 4 weeks
Drug: Dolormin® extra (Ibuprofen) — Ibuprofen Tablets (as lysine-salt) 2400mg/d (400mg 2-2-2) applied orally for 12 weeks (Arm II, n=6).
  In order to reduce the risk of damage to the gastrointestinal mucosa Pantoprazole is applied as concomitant medication in a dosage 40mg/d during the first 4 weeks of treatment and may be reduced to 20mg/d during the following treatment period after individual risk-benefit assessment.
  Other Names: Ibuprofen-DL-Lysinsalz
  Arms: Dolormin® extra (Ibuprofen) 12 weeks

SUMMARY:
The Ibuprofen - Spinal Cord Injury (SCI) - Safety trial investigates tolerability and feasibility of "small molecule" (Ibuprofen) mediated Rho-inhibition as putative neuroprotective, plasticity-enhancing and neurorestaurative intervention. The primary safety analysis is based on the incidence of severe gastrointestinal bleedings. In addition, the feasibility of recruitment procedure, and oral administration of the compound within the multidisciplinary setting of acute intensive medical care will be explored. Furthermore, the pharmacokinetics of Ibuprofen under the condition of acute motor complete SCI will be investigated. Secondary endpoints will permit preliminary statements about effects on neuropathic pain, spasticity, and neurological function.

ELIGIBILITY:
Inclusion Criteria:

* Acute SCI of the cervical spine due to trauma
* Time frame of 4-21 days post-trauma
* Motor complete injury AIS A and B
* Neurological level of the lesion C4-T4
* No participation in a different clinical trial according to German Pharmaceuticals Act (AMG) 1 month before and during participation in the current trial
* The patient has been informed and his/her written consent has been obtained
* Age: 18 to 65 years
* For women of reproductive age: Negative pregnancy test and highly effective contraception (defined as Pearl Index < 1) or sexual abstinence during participation in the trial

Exclusion Criteria:

* Multifocal lesions of the spinal cord
* Penetrating spinal cord injury
* Accompanying traumatic brain injury (TBI) with visible structural lesions including intracranial hemorrhage on diagnostic imagesSigni
* Significant accompanying injury to the peripheral nervous system, particularly plexus lesions
* Acute or chronic systemic diseases accompanied by neurological deficits or that have caused permanent neurological deficits which may overlay or hinder the registration of sensomotor functions (e.g. multiple sclerosis, Guillain-Barré syndrome, HIV infection, Lues etc.)
* Malignant neoplasms, except if these are in complete remission.
* Mental diseases or dementia which, in the investigator's opinion, limit the patient's cooperation in respect of the intake of the study medication and/or significantly hinder the registration of follow-up parameters
* Hemophilia
* History of myocardial infarction or stroke
* Current and persistent misuse of illegal drugs or alcohol
* Hypothermia below 35 C°
* Pregnancy and lactation
* All further contraindications to the study medication, including other ingredients of the pharmaceutical form according to the Summary of Product Characteristics (SPC)
* Known hypersensitivity to the active substance contained in the concomitant medication Pantoprazole or one of the components of the drug.
* Intake of Ibuprofen or intake of other active substances from the group of Nonsteroidal Anti-inflammatory Drugs (NSAIDs; e.g., Diclofenac, Indometacin) or the intake of NSAIDs in maximum recommended daily doses during one week prior to enrolment in the trial
* Simultaneous intake of salicylates, particularly acetylsalicylic acid
* Simultaneous intake of oral anticoagulants
* Simultaneous intake of systemic glucocorticoids
* Unwilling to consent to storage and transfer of pseudonymized medical data for the purpose of the clinical trial
* Admitted to an institution by a court or official order (pursuant to AMG §40 (1) 4)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with severe gastroduodenal bleedings as a measure of safety | up to 4 months
  Safety of lbuprofen as measured by the occurence of severe gastroduodenal bleedings documented as serious adverse events (SAE)

SECONDARY OUTCOMES:
Spasticity on the Modified Ashworth Scale (MAS) | 4 weeks and 6 months
Pain on the Neuropathic Pain Scale (NPS) | baseline, 4 weeks and 6 months
International standards for neurological classification of spinal cord injury (ISNCSCI) - ASIA impairment scale (AIS) change from baseline | baseline, 4 weeks and 6 months
Neurological motor function on the ISNCSCI/ASIA motor scores change from baseline | baseline, 4 weeks and 6 months
Neurological sensory function on the ISNCSCI/ASIA sensory score change from baseline | baseline, 4 weeks and 6 months
Number of participants with adverse events as a measure of safety and tolerability | up to 6 months
Ibuprofen levels in plasma | Arm I (day 1 and week 4), Arm II (day 1, week 4 and 12) 1.5 and 3 hours post-dose
Ibuprofen levels in cerebrospinal fluid (CSF) | Arm I (day 1 and week 4), Arm II (day 1, week 4 and 12) 3 hours post-dose

OTHER OUTCOMES:
Heterotopic ossifications | baseline, 4 weeks and 6 months
  Screening for heterotopic ossifications using sonography of the hip joints

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Niedeggen, MD, Principal Investigator — Unfallkrankenhaus Berlin, Treatment Centre for Spinal Cord Injuries, Germany; Jan M Schwab, MD, PhD, Study Director — Charité, Universitätsmedizin Berlin, Spinal Cord Injury Research, Germany
Locations (1):
- Unfallkrankenhaus Berlin, Treatment Centre for Spinal Cord Injuries, Warener Straße 7, Berlin, Germany

REFERENCES:
- [Derived] Kopp MA, Liebscher T, Watzlawick R, Martus P, Laufer S, Blex C, Schindler R, Jungehulsing GJ, Knuppel S, Kreutztrager M, Ekkernkamp A, Dirnagl U, Strittmatter SM, Niedeggen A, Schwab JM. SCISSOR-Spinal Cord Injury Study on Small molecule-derived Rho inhibition: a clinical study protocol. BMJ Open. 2016 Jul 26;6(7):e010651. doi: 10.1136/bmjopen-2015-010651. PMID 27466236